CLINICAL TRIAL: NCT04392830
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study, to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses (SAD-MAD) of ALZ002 DS in Healthy Volunteers
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics of ALZ002 DS in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnnJi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ALZ002-101
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALZ002 DS (Experimental): SAD: 6 cohorts of subjects are planned to be orally dosed, ranging from 15 mg - 800 mg.
  MAD: 3 cohorts of subjects are planned to be orally dosed once or twice daily for 7 consecutive days, ranging from 300 mg - 600 mg.
  Interventions: Drug: ALZ002 DS
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALZ002 DS — Administered orally
  Other Names: JM17
  Arms: ALZ002 DS
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of single-ascending and multiple-ascending doses of ALZ002 DS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or non-childbearing potential female subjects, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤55 years of age at screening.
* Body mass index > 18.5 and < 30.0 kg/m2, and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females at screening visit.
* Capable of consent.

Exclusion Criteria:

* Any clinically significant abnormality or abnormal laboratory test results
* Positive urine drug screen, alcohol breath test, or urine cotinine test
* History of significant allergic reactions to any drug.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device
* History of clinically significant opportunistic infection
* Presence of fever (body temperature > 38°C)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of SAEs and treatment-related adverse events | Baseline through Study Completion (up to Day 14)
  Incidence of SAEs and treatment-related severe AEs

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) will be assessed | predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose; Day 3: predose; Day 4:predose; Day 5:predose; Day 6: predose; Day7: predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose
  Maximum observed plasma concentration (Cmax)
Area Under the Curve (AUC) will be assessed | predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose; Day 3: predose; Day 4:predose; Day 5:predose; Day 6: predose; Day7: predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose
  Area under the plasma concentration versus time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Cmax clinical research, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No